CLINICAL TRIAL: NCT06902610
Title: Observational Follow-up Study Examining the Medium-term Effect on Non-inferiority of the Previous Training With the Digital Medical Device (DMD) Poppins Clinical for Cognitive and Musical Training in Addition to Bi-monthly Speech and Reading Therapy Sessions on the Reading and Writing Abilities of Pediatric Patients With Specific Learning Disorders Involving Reading and/or Writing Deficits (SLD Reading) Compared to a Control Group Receiving Weekly Speech and Reading Therapy Sessions (POPPINS-02-b, Ancillary Study to POPPINS-02)
Brief Title: Examining the Medium-term Effect on Non Inferiority of the Previous Training With the DMD Poppins Clinical for Cognitive, Musical Training in Addition to Bi-monthly Speech and Reading Therapy on Reading Writing Abilities of Pediatric Patients With SLD Reading VS Control Group
Acronym: POPPINS-02-B
Status: Recruiting | Type: Observational
Sponsor: Poppins (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Other Study IDs: POPPINS-02-b
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Learning Disorder, Specific; Learning Disability; Specific Learning Disorder, With Impairment in Reading; Dyslexia
MeSH Terms: conditions — Specific Learning Disorder; Learning Disabilities; Dyslexia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No intervention: CONTROL: 1 session of speech and reading therapy weekly, no use of the medical device Poppins Clinical
- Experimental: Reduced speech and reading therapy sessions (1 session every 2 weeks) and use of the medical device Poppins Clinical
  Interventions: Device: Poppins Clinical

INTERVENTIONS:
Device: Poppins Clinical — Poppins Clinical is a software as a medical device that combines a musical and combines a musical and cognitive training program and written language training program.
  Groups: Experimental

SUMMARY:
Poppins-02-b is an observational follow-up study examining the medium-term effect on non-inferiority of the previous training with the digital medical device (DMN) Poppins Clinical for cognitive and musical training in addition to bi-monthly speech and reading therapy sessions on the reading and writing abilities of pediatrics patients with specific learning disorders involving reading and/or writing deficits compared to a control group that received weekly speech and reading therapy sessions.

Poppins-02-b is an ancillary study to Poppins-02 and consists of monitoring patients who participated in Poppins-02 study.

DETAILED DESCRIPTION:
The POPPINS-02-b follow-up study consists in following up patients who took part in the POPPINS-02 clinical trial: a randomized non-inferiority trial with a control group designed to assess the effect of adding the Poppins Clinical digital medical device in addition to bi-monthly speech and reading therapy sessions on the skills of patients with reading disorders. Patients included in the original POPPINS-02 study were randomized into one of two groups:

1. Experimental group (EXPE group): will receive the Poppins Clinical digital medical device in addition to bi-monthly speech and reading therapy sessions.
2. Control group (CONT group): will receive weekly speech and reading therapy sessions.

In the original POPPINS-02 study, the experimental phase lasts 12 weeks in total, with a preliminary evaluation (T1) and a final evaluation (T2) after this period.

All patients enrolled in the POPPINS-02 study will be included, if they so wish, in the POPPINS-02-b follow-up study. This study consists of a 12-week follow-up phase after the final POPPINS-02 protocol visit (T2). During this follow-up phase, all patients will return to their usual speech therapy management with the frequency planned before their participation in POPPINS-02. During this follow-up phase, patients in both groups will not have access to the Poppins Clinical application. At the end of the 12-week follow-up period, an evaluation (T3) is scheduled. Assessments will cover primary, secondary and exploratory endpoints.

A questionnaire will also be submitted to parents and speech therapists caring for the children during T3 in order to collect information on the dates of speech therapy sessions during this follow-up period, and to benefit from their perspective on the medium-term effect of the study protocol on speech therapy follow-up.

Access to the Poppins Clinical digital medical device will be offered to children in the two POPPINS-02 study groups who decide to participate in the POPPINS-02-b follow-up study at the end of the experiment.

The investigator and his team will remain blind as to which groups will be assigned to the POPPINS-02 study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria:
* Patient who has been enrolled in the POPPINS-02 study.
* Participation agreement from the patient as well as from the legal guardians, and commitment to follow the protocol.

Exclusion Criteria:

* Any pathology that, at the discretion of the investigator, may prevent the patient from participating in the study.
* Patient participating in an interventional study that could affect the results.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: According to the DSM-5-TR or ICD-11 Specific Learning Disability (SLD) or Developmental Learning Disability (DLD) is one of the most common neurodevelopmental disorders. It affects between 5% and 15% of schoolchildren. In particular, SLD is one of the most common neurodevelopmental disorders. It affects between 6% and 8% of schoolchildren. It is characterized by significant and persistent difficulties in the acquisition of academic skills, which may include reading, writing or arithmetic, although dyslexia is by far the most common type, accounting for 80% of SLD. SLD first manifests itself during the teaching of academic or occupational functioning. Children with SLD do not have associated intellectual retardation, overt brain damage or degenerative disorders. They are therefore likely to benefit most from remediation.
Sampling Method: Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the medium term non-inferiority of Poppins Clinical as a complement to reduced speech and reading therapy compared to only speech and reading therapy | 12 weeks
  This endpoint evaluates the non-inferiority on reading abilities using a word reading task measured by the 2-minutes word reading rest form EVALEO (EVAL2M), assessing the number of words correctly read, 12 weeks after the last evaluation of the POPPINS-02 study

SECONDARY OUTCOMES:
Evaluate the medium-term effect of adding Poppins Clinical on reading abilities (in terms of reading speed) (non-inferiority). | 12 weeks
  This endpoint evaluates the non-inferiority on reading abilities using a word reading task measured by the 2-minute word reading test from EVALEO (EVAL2M), assessing the number of words read, 12 weeks after the last evaluation of the POPPINS-02 study.
Evaluate the medium-term effect of adding Poppins Clinical on text reading skills (non-inferiority). | 12 weeks
  This endpoint evaluates the mid-term effect of the addition of Poppins Clinical on word reading skills in terms of speed and accuracy as assessed by a text reading test (Alouette) (speed and accuracy scores), 12 weeks after the last evaluation of the POPPINS-02 study.
Assessment of the medium-term effect of adding Poppins Clinical on parental stress level between the two groups (EXP/CONT) (non-inferiority). | 12 weeks
  This endpoint examines the mid-term impact of adding Poppins Clinical on parents' stress levels, measured using the parenting stress index short form, 12 weeks after the last evaluation of the POPPINS-02 study.
Description and comparison of the medium-term effect of adding Poppins Clinical on the quality of life of parents between the two groups (EXP/CONT) (non-inferiority). | 12 weeks
  This endpoint examines the mid-term impact of adding Poppins Clinical on parents' quality of life, measured using the EQ-5D-5L quality of life questionnaire, 12 weeks after the last evaluation of the POPPINS-02 study.
Evaluate the medium-term effect of adding Poppins Clinical on metaphonological skills (non-inferiority). | 12 weeks
  This endpoint evaluates the mid-term effect of adding Poppins Clinical on meta-phonological skills as assessed by the BALE phoneme suppression test (correct answers score), 12 weeks after the last evaluation of the POPPINS-02 study.
Evaluate the medium-term effect of adding Poppins Clinical on text comprehension (non-inferiority). | 12 weeks
  This endpoint evaluates at the mid-term effect of adding Poppins Clinical on text comprehension assessed using the computerized adaptable test battery (BMT-i) (evaluated scores: correct answers to text comprehension questions score, reading precision and speed), 12 weeks after the last evaluation of the POPPINS-02 study.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Henri Laborit, Poitiers

IPD SHARING:
Plan to Share IPD: No